CLINICAL TRIAL: NCT06896656
Title: Improving Social Connectedness Through Digital Health to Enhance Recovery from OUD Among the Justice Involved Population
Acronym: STAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34DA058299 (NIH)
Record Dates: First submitted 2025-03-12; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Loneliness; Opioid Use Disorder
Keywords: Mobile Health
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Health Resources

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MPS App (Experimental): This is the experimental arm. Participants assigned to this arm will receive access to the Marigold Health App (MPS) intervention. N = 60 participants will be assigned to this arm.
  Interventions: Behavioral: Marigold Mobile Peer Support Intervention
- Enhanced Treatment as Usual (Active Comparator): This is the active comparator arm. Participants assigned to this arm will receive enhanced treatment as usual. N = 30 participants will be assigned to this arm.
  Interventions: Behavioral: Resources

INTERVENTIONS:
Behavioral: Marigold Mobile Peer Support Intervention — The MPS App is a secure platform that allows text-based peer support for individuals in recovery from OUD. Participants assigned to this condition will be enrolled on a rolling basis into a peer support group on the app. All participants will receive onboarding assistance and will have access to the app for 6 months.
  The app will include live moderation from a certified Peer Recovery Support Specialist and trained research assistants. Moderators will begin discussions with prompts and regulate the flow of conversation with standardized text language. Moderators will be able to respond in real-time to malicious messages or other "flags" that could impact participant safety. Built in natural language processing algorithms will also detect language requiring intervention and automatically alter the moderators and on-call clinicians.
  Arms: MPS App
Behavioral: Resources — A list of online peer support and mental health resources, drawn from SAMSHA and equivalent websites, will be provided to all participants, as an enhanced adjunct to their standard recovery plans.
  Arms: Enhanced Treatment as Usual

SUMMARY:
People with a history of Opioid Use Disorder and criminal justice involvement are more likely to experience loneliness following release from jail/prison leading to negative outcomes such as treatment dropout and increased substance use. Providing peer recovery support, particularly through a highly accessible, digital health platform, is a potential way to decrease loneliness in this population. The current study seeks to test whether a mobile peer recovery support app, delivered to individuals with a recent history of taking medication for opioid use disorder while in jail/prison, will improve outcomes for this vulnerable population.

DETAILED DESCRIPTION:
Individuals with criminal justice involvement experience elevated rates of Opioid Use Disorder (OUD) and are at significantly higher risk of death from opioid overdose in the first year following release from jail/prison. Medications for OUD (MOUD) are an evidence-based approach to treating OUD and offer extensive benefits including lowering rates of mortality, illicit opioid use, HIV transmission, violent crime, and arrest. While many correctional settings have started to implement MOUD, there are significant challenges to continuing medication/treatment while transitioning back to the community. Intersectional stigma related to addiction and history of incarceration is associated with greater difficulties with reintegration, increased isolation, and heightened feelings of loneliness. Lack of social connectedness further serves as a risk factor for decreased retention in treatment, discontinuation of MOUD, and a return to substance use. Peer support is a key component of many evidence-based OUD recovery programs. When used in conjunction with MOUD, it has the potential to improve perceived social support, self-efficacy, and treatment engagement. However, access to live peer support has been challenged by COVID restrictions, highlighting a critical need for digital health platforms to deliver peer support. The Marigold Mobile Peer Support ("MPS") App is a dedicated, secure, mobile application that employs structured, live peer moderation to guide text-based conversations with groups of participants and behind-the-scenes natural language processing (NLP) to automatically identify "red flag" content within peer chats. While initial work demonstrates the utility of deploying the MPS App in outpatient treatment settings for OUD, it has yet to be tested in correctional settings or among justice-involved populations. The goal of the proposed application is to advance evidence-based and scalable treatments for OUD, by decreasing loneliness and enhancing perceived social support via novel application of an established mobile app among individuals with a history of engaging in MOUD while in jail/prison. The study will be accomplished through two primary aims: (1) develop an implementation manual to guide delivery of the MPS App for those with a recent (past year) history of engaging in MOUD while in jail/prison by conducting in-depth interviews with prospective app users and other key stakeholders; and (2) conduct a randomized controlled trial to assess feasibility, acceptability, and preliminary efficacy of the MPS App relative to enhanced treatment-as-usual among individuals with a recent (past year) history of engaging in MOUD while in jail/prison. Findings from this study will be used to develop a R01 application to conduct a fully-powered Hybrid Type 1 Effectiveness-Implementation study.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* history of being prescribed medication for opioid use disorder (MOUD) while in jail or prison
* most recently released from prison with the past two years
* self-reported recovery for an Opioid Use Disorder (OUD)
* able to understand and speak English and to provide written and verbal consent
* anticipated discharge from jail/prison within 3 months if currently incarcerated

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Social Support | Baseline, 1, 3, and 6 months.
  Perceived social support will be assessed with the Multidimensional Scale of Perceived Social Support (MSPSS). This assessment is psychometrically sound, with adequate reliability and validity, and measures perceived social support from family, friends, and significant others among adults. Scores are averaged and range from 1 to 7, with 1 signifying the lowest level of social support and 7 signifying the highest.
Loneliness | Baseline, 1, 3, and 6 months.
  Loneliness will be assessed with the 20-item UCLA Loneliness scale. Scores range from 20 to 80, where higher scores indicate greater loneliness.

SECONDARY OUTCOMES:
Substance Use | Baseline, 1, 3, and 6 months.
  Self-reported substance use will be assessed with the Timeline Follow-Back interview and biochemically confirmed with Urine Drug Screens. Substance use will be operationalized as the percentage of days positive for drug use (separate by drug class) in between assessments.
Engagement in Medications for Opioid Use Disorder (MOUD) | Baseline, 1, 3, and 6 months.
  Self-reported engagement in MOUD will be assessed with a Timeline Follow-Back interview and biochemically confirmed with Urine Drug Screens. Engagement in MOUD will be operationalized as the percentage of days positive for MOUD administration in between assessments.

OTHER OUTCOMES:
Demographics | Baseline
  Using the PhenX toolkit, basic demographic data and social determinants of health will be collected. In addition, prior and current history with the criminal justice system will be assessed with the Adult Incarceration Module of the National Survey on Drug Use and Health (NSDUH) 2014 Questionnaire.
Treatment Received | Baseline, 1, 3, and 6 months.
  The Treatment Services Review will be administered to assess receipt of case management, psychiatric, peer recovery coaching, and other treatment services, including utilization of MOUD. At follow-up interviews, participants will be asked about the services received since the previous interview.
Quality of Life | Baseline, 1, 3, and 6 months.
  The Quality of Life Enjoyment and Satisfaction Questionnaire Short Form, a 16-item questionnaire with sound psychometric properties, will be administered to assess quality of life. Scores range from 0 to 100, with higher scores indicating greater enjoyment and satisfaction.
Wellbeing | Baseline, 1, 3, and 6 months.
  The World Health Organization-Five Well-Being Index (WHO-5) will be administered to assess wellbeing. This 5-item questionnaire is a widely used and valid tool for assessing wellbeing. Scores range from 0 to 100, with 0 representing the worst possible wellbeing and 100 representing the best possible wellbeing.
Depressive Symptoms | Baseline, 1, 3, and 6 months.
  Depressive symptoms will be assessed with the Patient Health Questionnaire-2 (PHQ-2). This measure consists of 2 items with high sensitivity, specificity, and discriminant validity for diagnosing major depression. Scores range from 0 to 6. A score of 3 or greater indicates major depression disorder is likely.
Anxiety Symptoms | Baseline, 1, 3, and 6 months.
  Anxiety symptoms will be assessed with the Generalized Anxiety Disorder 2-Item (GAD-2). This measure consists of 2 items and has well established accuracy for identifying clinically significant anxiety symptoms and tracking treatment progress outcomes. Scores range from 0 to 6. A score of 3 or greater indicates a high likelihood of generalized anxiety disorder diagnosis.
Perceived Stress | Baseline, 1, 3, and 6 months.
  The Perceived Stress Scale (PSS-10) will be administered to assess perceived stress in the past month. The PSS-10 consists of 10 items and is psychometrically sound. Scores range from 0 to 40, with 40 representing the highest possible perceived stress.
Number of Days of App Use | 6 months
  The number of days participants use the Marigold Health app will be extracted from the app as indices of app engagement.
Number of Messages Sent in App | 6 months
  The number of messages a participant sends in the Marigold Health app will be extracted from the app as an indices of app engagement.
System Usability Scale | 6 months
  The System Usability Scale will be administered to participants in the treatment arm. This assessment measures perceived usability of digital systems. Scores range from 0 to 100, with 100 representing high perceived usability. These scores will be used as indices of app satisfaction.
Client Satisfaction Questionnaire | 6 months
  The Client Satisfaction Questionnaire will be administered to participants in the treatment arm. This measure of intervention satisfaction consists of 8 items. Scores range from 8 to 32, with higher scores indicting higher satisfaction. These scores will serve as indices of app satisfaction.
Qualitative Exit Interview | 6 months
  Qualitative exit interviews will be conducted with a subset of participants (n = 20) assigned to the treatment arm. The interviews will be used to collect in-depth feedback about the intervention.
Number of Flagged Messages | 6 months
  The number of messages flagged in the Marigold Health app will be extracted from the app. This will serve as indices of safety of the app.
Number of Crisis Interventions | 6 months
  The number of crisis interventions clinicians administer to participants using the Marigold Health app will be extracted from the app. This will serve as indices of app safety.
Time Spent Onboarding App Users | 6 months
  The amount of time required for research staff to onboard users to the Marigold Health app will be recorded. This will serve as indices of intervention scalability.
Clinician Time Spent on Crisis Managment | 6 months
  The amount of time it takes clinicians to manage emergent crises on the Marigold Health app will be recorded. This will serve as indices of intervention scalability.

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No